CLINICAL TRIAL: NCT00454064
Title: Study to Compare a Cognitive-behavioral Treatment With a Cognitive-behavioral Treatment With Biofeedback Elements to Patients With Chronic (Low) Back Pain
Brief Title: Cognitive-behavioural Treatment of Chronic Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGT090774
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Back Pain
Keywords: cognitive-behavioral therapy; back pain; low back pain; biofeedback; randomized controlled study; EMG biofeedback
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): cognitive-behavioral treatment
  Interventions: Behavioral: cognitive-behavioral treatment
- 2 (Active Comparator): cognitive-behavioral treatment with biofeedback elements
  Interventions: Behavioral: cognitive-behavioral treatment

INTERVENTIONS:
Behavioral: cognitive-behavioral treatment

SUMMARY:
The purpose of the study:

* to compare two cognitive-behavioral treatments

DETAILED DESCRIPTION:
128 patients suffering from chronic back pain were randomly assigned to either Wait List Control, Cognitive Behavioral Treatment or Cognitive Behavioral Treatment and Biofeedback.

Measures were conducted 6 months before treatment (Wait List Control) immediately before and after treatment and at 6-months follow-up.

25 weekly 1-hr sessions of individualized outpatient cognitive behavioral treatment of chronic back pain

Treatment elements:

Cognitive treatment: identification, evaluation and correction of dysfunctional beliefs about themselves and pain by cognitive restructuring, problem-solving training and coping skills training

Behavioural treatment: increasing activity levels (sports, social activities, work), reducing medication intake and unnecessary health care utilization Relaxation training: progressive muscle relaxation, biofeedback.

ELIGIBILITY:
Inclusion Criteria:

* Back pain since 6 months

Exclusion Criteria:

* Patients with psychosis, borderline psychopathy, drug dependence i.e. alcohol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
pain intensity | start of treatment, end of treatment, 6-months follow-up

SECONDARY OUTCOMES:
pain disability | start of treatment, end of treatment, 6-months follow-up
depression | start of treatment, end of treatment, 6-months folow-up

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Professor, Study Chair — University Marburg, Department of Clinical Psychology and Psychotherapy
Locations (1):
- University Marburg, Department of Clinical Psychology and Psychotherapy, Marburg, Hesse, Germany